CLINICAL TRIAL: NCT06709742
Title: Effect of Goal-Oriented GMFM-88 Based Program on Enhancing Gross Motor Function, Balance and Quality of Life Among Children with Cerebral Palsy
Brief Title: Effect of Goal-Oriented GMFM-88 Based Program in Cerebral Palsy.
Acronym: CP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Ifra Neelum, Principle Investigator, Ziauddin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 8750524INREH
Record Dates: First submitted 2024-11-18; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Palsy; Quality of Life (QOL); Balance; CP
Keywords: Cerebral Palsy; Gross motor function; Balance; Quality of Life; CP; GMFM-88; BESTest; CP QOL
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental): The Intervention based on GMFM-88 items will be given 3 times per week for a duration of 40-45 minutes for each session for 16 weeks.
  Interventions: Other: Gross Motor Function Measure-88 Based Therapy

INTERVENTIONS:
Other: Gross Motor Function Measure-88 Based Therapy — Children will be assessed initially by using GMFM-88 and selecting specific items for individuals according to his/her needs with the help of experts and family. At least 3 items will be selected for each subject in which they score less such that 0, 1 or 2. Training based on those specific items will be given to the children. This is goal-oriented training in which, according to the needs of children training will be provided.
  Other Names: GMFM-88 Based Therapy

SUMMARY:
Cerebral Palsy (CP) is a infancy and early childhood disorder that results in motor impairment caused by static and non-progressive lesions in the brain. It has an impact on both the neurological and musculoskeletal systems of the bod. According to the Cerebral Palsy Alliance Research Foundation (CPARF) & WHO Cerebral Palsy Statistics 2023, approximately 17 million individuals experience some form of CP. This data underscores a notable prevalence rate of 1.5 cases per 1,000 live births within the High-Income Countries (HICs), limited but growing data are obtained from both the Lower Middle-Income Countries (LMICs. The incidence of CP among children in the Swabi district of Khyber Pakhtunkhwa, Pakistan, was 1.22 per 1000 live births. The overall prevalence in Pakistan is still not known, but according to recent documentation, it is estimated to be 4 out of every 1000 live births.

The symptoms in CP encompassing atypical muscle contractions, alteration in posture and limitations in movement and physical activity. Furthermore,these symptoms are accompanied by disruptions in sensory perception and cognitive processing along with the challenges of communication, behavioral issues, epileptic seizures and secondary musculoskeletal complications. Motor deficit is present in 65.56% percent of CP cases as well as balance is impaired in most of the cases, and different impairments combinedly decreased overall quality of life (QOL). Because activities of daily living are decreased which in a result increases the caregiver's workload.Despite such a high prevalence of CP, there is still no standardized treatment approach implemented in the clinical settings due to their individualized needs and varying degrees of impairment.

Consequently, our study seeks to address this gap by investigating the effect of Goal-Oriented individualized GMFM based programs on enhancing gross motor function, balance and quality of life. By elucidating the potential benefits of intervention, our study aims to contribute to the optimization of therapeutic approaches tailored to the different needs of children with CP.

DETAILED DESCRIPTION:
A total number of 47 participants will be included in the study. A written informed assent will be taken from the parent or guardian of the child prior to intervention which includes a detailed description of the method, procedure, benefits and risks of the training. Children will perform GMFM-88 based individualized goal-oriented training selected with the concern of family and caregivers. All children will be assessed initially based on GMFCS level and categorized into levels I, II & III. Baseline assessment will be carried out before the first session of all the recruited children using GMFM-88 to assess gross motor function, Kids-Balance Evaluation-System (Kids-BESTest) for balance & Quality of Life assessed through CPQOL questionnaire respectively. Children will be reassessed after the 16 weeks of training and re-evaluated on the 18th for residual effects after completion of 16 weeks of training. The intervention will be given 3 times per week for a duration of 40-45 minutes for each session for 16 weeks (In addition, a written home program will be given to the parents/guardians of the participants to carry out the program at home). To ensure that the parents are regularly performing exercises a WhatsApp group will be created for sending reminders. Parents will be appreciated and motivated through messages. After completing the home program parents will send a message.

Goal Oriented Exercise Protocol:

After screening the children will perform GMFM-88 based goal-oriented training assigned by trained therapists such as items of dimension D are related to standing and dimension E items are related to walking and running. 5-10 minutes of warm-up provided preliminary. Including stretching, bridging, upper and lower limb range of motions. Children will be assessed initially by using GMFM-88 and selecting specific items for individuals according to his/her needs with the help of experts and family. At least 3 items will be selected for each subject in which they score less such that 0, 1 or 2. Training based on those specific items will be given to the children. This is goal-oriented training in which, according to the needs of children training will be provided. There are 13 items in dimension D and 24 items in dimension E. At the end of the study, we analyze the children's number on each item and their improvement after the training.

Dimension D: Standing Items of dimension included such as maintaining standing with and without arms, lifting a single leg from the floor, sitting to stand, attaining standing from high kneeling, squats and picking objects from the floor.

Dimension E: Walking, Running & Jumping

Dimension E included items such as cruising, forward and backward walking, turning 180 degrees, walking on parallel and straight lines, crossing hurdles, running, kicking ball, jumping, hopping, ascending and descending stairs.MATCHING ACTIVITIES:

1. DIMENSION D (STANDING):

   * The child stands with the wall support at the back and engages in catch and throw activities with his peers/therapist.
   * The child stands against the wall with a table in front to be engaged in the activity.
   * The child is asked to kick the ball with/without holding a parallel bar.
   * For one leg standing balance, the child's one leg will be placed on the football while the other on the floor.
   * Placing alternate feet on the bench of 0.5 feet in height.
   * Sit to stand from the 1-foot high bench, a key point of control /assistance as needed.
2. DIMENSION E (WALKING & RUNNING):

   * Walking holding onto the parallel bar.
   * Walking while holding a book/toy in hand.
   * Motivate the child to climb up and down stairs starting with rail support and progressing to without rail support. Initially with both feet and then progress to a single foot.
   * Cruising on the left and right side using furniture for support.
   * Crossing over the small obstacles of varying height (child's ankle, mid calf & knee level).
   * Making figures of 8 while walking.
   * Jumping on the same mark.
   * Hold the parallel bar with hand and kick the ball.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosed Cerebral Palsy,

  * Age 5-16 years,
  * GMFCS Level I, II & III,
  * Able to understand instructions,
  * With/ without any assistive devices.

Exclusion Criteria:

* • CP children with any respiratory disorders,

  * Undergoing surgery within the past 6 months,
  * Botulinum injection within the last 6 months,
  * Unstable seizures,
  * Co-existing condition (ADHD, Metabolic Disorder, Progressive disorder),
  * Any other co-morbid causing difficulty in performing tasks.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function | At Baseline
  The GMFM-88 (Gross Motor Function Measure-88) is a scale used to assess gross motor function in children with CP.
Gross Motor Function | Through study completion, at 16th week
  The GMFM-88 (Gross Motor Function Measure-88) is a scale used to assess gross motor function in children with CP.
Gross Motor Function | followup of 2 weeks.
  The GMFM-88 (Gross Motor Function Measure-88) is a scale used to assess gross motor function in children with CP.
Balance | At Baseline
  The Kids BESTest Scale (Balance Evaluation Systems Test) is used to assess balance in children with CP.
Balance | Through study completion, at 16th week
  The Kids BESTest Scale (Balance Evaluation Systems Test) is used to assess balance in children with CP.
Balance | followup of 2 weeks.
  The Kids BESTest Scale (Balance Evaluation Systems Test) is used to assess balance in children with CP.
Quality Of Life | At Baseline
  The CP QOL (Cerebral Palsy Quality of Life) questionnaire is used to assess the quality of life in children with CP.
Quality Of Life | Through study completion, at 16th week
  The CP QOL (Cerebral Palsy Quality of Life) questionnaire is used to assess the quality of life in children with CP.
Quality Of Life | followup of 2 weeks.
  The CP QOL (Cerebral Palsy Quality of Life) questionnaire is used to assess the quality of life in children with CP.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Amna Aamir Khan, PhD, Study Director — Ziauddin College of Physical Therapy, Ziauddin University; Ifra Neelum, MPhil, Principal Investigator — Ziauddin College of Physical Therapy, Ziauddin University
Locations (2):
- Pakistan (2):
  - ACELP Institute of Child Development, Karachi, Sindh
  - Dar-ul-Sukun, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee M, Ko Y, Shin MM, Lee W. The effects of progressive functional training on lower limb muscle architecture and motor function in children with spastic cerebral palsy. J Phys Ther Sci. 2015 May;27(5):1581-4. doi: 10.1589/jpts.27.1581. Epub 2015 May 26. PMID 26157267
- [Background] Paul S, Nahar A, Bhagawati M, Kunwar AJ. A Review on Recent Advances of Cerebral Palsy. Oxid Med Cell Longev. 2022 Jul 30;2022:2622310. doi: 10.1155/2022/2622310. eCollection 2022. PMID 35941906
- [Background] McIntyre S, Goldsmith S, Webb A, Ehlinger V, Hollung SJ, McConnell K, Arnaud C, Smithers-Sheedy H, Oskoui M, Khandaker G, Himmelmann K; Global CP Prevalence Group*. Global prevalence of cerebral palsy: A systematic analysis. Dev Med Child Neurol. 2022 Dec;64(12):1494-1506. doi: 10.1111/dmcn.15346. Epub 2022 Aug 11. PMID 35952356
- [Background] Cooper MS, Fahey MC, Mackay MT. Making waves: The changing tide of cerebral palsy. J Paediatr Child Health. 2022 Nov;58(11):1929-1934. doi: 10.1111/jpc.16186. Epub 2022 Sep 6. PMID 36066306
- [Background] Abd-Elfattah HM, Ameen FH, Elkalla RA, Aly SM, Abd-Elrahman NAF. Loaded Functional Strength Training versus Traditional Physical Therapy on Hip and Knee Extensors Strength and Function Walking Capacity in Children with Hemiplegic Cerebral Palsy: Randomized Comparative Study. Children (Basel). 2022 Jun 24;9(7):946. doi: 10.3390/children9070946. PMID 35883930